CLINICAL TRIAL: NCT00451243
Title: Differential Clinical and Serologic Response in Psoriasis and Psoriatic Arthritis to Drug Treatmen
Brief Title: Differential Clinical and Serologic Response in Psoriasis and Psoriatic Arthritis to Drug Treatment
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701244; 9361701244
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2004-12

CONDITIONS: Psoriatic Arthritis
Keywords: psoriatic arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Psoriasis is a multifactorial cutaneous disorders which affects about 100000 patients in Taiwan. Psoriatic arthritis is also present in about 20~30 percents. Many drugs have been shown to aggravate psoriasis including drugs used in the treatment of psoriatic arthritis. On the contrary, anti-psoriatic drugs are also known to aggravate or induce psoriatic arthritis. Psoriasis and psoriatic arthritis are believed to share the same pathogenic lymphocytes, but the differential responses to drugs are intriguing. This also causes problems in the treatment of psoriasis and psoriatic arthritis. Recently different serologic markers have been found for the assessment of psoriasis and psoriatic arthritis. Recent genetic study showed a different genetic susceptibility genes. We tested the serologic responses of three new biologic drugs used in the treatment of psoriasis and psoriatic arthritis. Paired blood samples of the same patients before and after 12 weeks of treatment were used. IL6 decreased after alefacept and etanercept but was increased after efalizumab treatment without statistical significance (Paired t test: 0.3336、0.2773、0.5904)。IL-8 decreased after etanercept but increased after efalizumab and alefacept without statistical significance (Paired t test: 0.4031、0.6749、0.2998)。IL10 decreased after efalizumab and etanercept, but increased significantly after alefacept treatment (Paired t test: 0.7254、0.5123、0.0350)。None of the treatment has a significant effect on TNF-alpha. HC10 decreased after alefacept and efalizumab,but increased after etanercept treatmentwithout statistical significance (Paired t test: 0.6589、0.1576、0.1988).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psoriasis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2005-01; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: TSEN-FANG Tsai, Study Chair — TSEN-FANG Tsai